CLINICAL TRIAL: NCT05432401
Title: Clinical Study of TAA05 Injection in the Treatment of Adult Patients With FLT3-positive Relapsed/Refractory Acute Myeloid Leukemia
Brief Title: TAA05 Injection in the Treatment of Adult Patients With FLT3-positive Relapsed/Refractory Acute Myeloid Leukemia
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: PersonGen BioTherapeutics (Suzhou) Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PG-pCART-TAA05-001
Record Dates: First submitted 2022-06-10; First posted 2022-06-27 (Actual); Last update posted 2022-06-27 (Actual); Status verified 2022-06

CONDITIONS: FLT3-positive Relapsed/Refractory Acute Myeloid Leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Acute

STUDY DESIGN:
Intervention Model Description: TAA05 Injection
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- T cell injection targeting FLT3 chimeric antigen receptor (Experimental): The subjects, who sign the informed consent forms and been screened by inclusion/exclusion criteria, will be assigned into 1.0 × 10^8, 2.0 × 10^8 and 4.0 × 10^8 CAR-T groups in order of sequence. And the subjects will be administered once.
  Interventions: Biological: T cell injection targeting FLT3 chimeric antigen receptor

INTERVENTIONS:
Biological: T cell injection targeting FLT3 chimeric antigen receptor — The subjects, who sign the informed consent forms and been screened by inclusion/exclusion criteria, will be assigned into 1.0 × 10^8, 2.0 × 10^8 and 4.0 × 10^8 CAR-T groups in order of sequence. And the subjects will be administered once.
  Other Names: TAA05 Injection

SUMMARY:
This is a single arm , open-label, dose-escalation clinical study with the primary objective of evaluating the safety and tolerability of TAA05 injection in adult subjects with FLT3-positive relapsed/refractory acute myeloid leukemia. The secondary objectives are as follows: to evaluate the in vivo expansion and persistence of FLT3-targeted chimeric antigen receptor T (CAR-T) cells after injection of TAA05;to evaluate the proportion of FLT3-positive cells in peripheral blood after injection of TAA05;to preliminarily evaluate the efficacy of TAA05 injection in adult subjects with FLT3-positive relapsed/refractory acute myeloid leukemia;to evaluate the immunogenicity of TAA05 injection;and to explore the applicable dose in the formal clinical phase.

DETAILED DESCRIPTION:
Approximately 1 sites are planned to be selected for the clinical trial. The subjects, who sign the informed consent forms and been screened by inclusion/exclusion criteria, will be assigned into 1.0 × 10^8, 2.0 × 10^8 and 4.0 × 10^8 CAR-T groups in order of sequence. And the subjects will be administered once. Dose escalation will follow 3 + 3 design and 3-6 subjects in each group will complete a single dose. Within the same dose group, the next subject will be administered after the previous subject has completed at least 14 days of safety observation. After the last subject in each dose group has completed the dose-limiting toxicity (DLT) assessment window of 28 days after single dose, the enrollment and treatment for the next dose group may be initiated after the Safety Review Committee (SRC) agrees to enter the next dose group based on clinical safety data assessment.

When DLT occurs in 1 of 3 subjects in a dose group, 3 additional subjects in the same dose group will be required (up to 6 subjects in the dose group have completed DLT assessment): if no DLT occurs in the additional 3 subjects, dose escalation will continue; if 1 of the 3 additional subjects experiences one DLT, dose escalation will be discontinued; if more than 1 of the 3 additional subjects experiences DLTs, dose escalation will be discontinued, and 3 additional subjects will be required to be enrolled at one lower dose level for DLT assessment. After the end of escalation for the maximum dose group, if no MTD is observed, the highest dose level is defined as the MTD.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 to 70 years old (inclusive), male or female;
* Expected survival time ≥ 3 months;
* ECOG performance status of 0-2;
* A clear diagnosis of acute myeloid leukemia at screening and positive expression of FLT3 in tumor cells;
* Subjects with relapsed/refractory acute myeloid leukemia who have failed standard treatment or lack effective treatment and meet any of the following criteria:

  1. After AML complete remission (CR), leukemia cells reappeared in peripheral blood or blast cells in bone marrow ≥ 5% (except for other reasons such as bone marrow regeneration after consolidation chemotherapy) or extramedullary leukemia cell infiltration;
  2. Initial cases that failed after 2 courses of standard treatment;
  3. After CR, patients with relapse within 12 months after consolidation and intensive treatment;
  4. Patients who relapsed after 12 months but did not respond to conventional chemotherapy;
  5. 2 or more relapses; persistent extramedullary leukemia;
* Coagulation function, liver and kidney function, cardiopulmonary function meet the following requirements:

  1. Prothrombin time/international normalized ratio (PT/INR) and partial thromboplastin time≤1.5 ULN;
  2. Creatinine≤1.5 ULN;
  3. Left ventricular ejection fraction≥50%, and no pericardial effusion was found on echocardiography, and no clinically significant abnormal bands were found on electrocardiography;
  4. Indoor baseline oxygen saturation>92%;
  5. Total bilirubin ≤ 2 × ULN; ALT and AST ≤ 2.5 × ULN; for ALT and AST abnormalities due to disease (e.g., liver infiltration or bile duct obstruction) as judged by the investigator, the indicators can be relaxed to ≤ 5 × ULN;
* Patients who can understand the trial and have signed informed consents.

Exclusion Criteria:

* Subjects with malignant tumors other than acute myeloid leukemia within 5 years prior to screening, with the exception of adequately treated cervical carcinoma in situ, basal cell carcinoma or squamous cell carcinoma, localized prostate cancer after radical surgery, and ductal carcinoma in situ after radical mastectomy;
* Positive for hepatitis B surface antigen (HBsAg) or hepatitis B core antibody (HBcAb) with peripheral blood hepatitis B virus (HBV) DNA titer detection not within the normal reference range; positive for hepatitis C virus (HCV) antibody and peripheral blood hepatitis C virus (HCV) RNA; positive for human immunodeficiency virus (HIV) antibody; positive for cytomegalovirus (CMV) DNA test; positive for syphilis test;
* Severe heart disease: including but not limited to unstable angina, myocardial infarction (within 6 months prior to screening), congestive heart failure (New York Heart Association [NYHA] classification ≥ III), severe arrhythmia;
* Unstable systemic diseases judged by the investigator: including but not limited to serious liver, kidney or metabolic diseases requiring drug treatment;
* Within 7 days prior to screening, there are active or uncontrollable infections requiring systemic therapy (except for mild genitourinary infection and upper respiratory tract infection);
* Pregnant or lactating women, and female subjects who plan to become pregnant within 2 years after cell infusion or male subjects whose partners plan to become pregnant within 2 years after cell infusion;
* Subjects who are receiving systemic steroid therapy within 7 days prior to screening or need long-term use of systemic steroid therapy during treatment as judged by the investigator (except for inhalation or topical use);
* Subjects who have participated in other clinical studies within 1 months prior to screening;
* Subjects who have evidence of central nervous system invasion at screening, such as tumor cells detected in cerebrospinal fluid or imaging suggesting central infiltration;
* Patients with graft-versus-host reaction and need to use immunosuppressants;
* Patients with a history of epilepsy or other central nervous system diseases;
* Patients with primary immunodeficiency disease;
* Conditions not eligible for cell preparation as judged by the investigator;
* Other conditions considered unsuitable for enrollment by the investigator.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2022-06-09 (Actual); Primary Completion 2023-06-09 (Estimated); Study Completion 2025-06-09 (Estimated)

PRIMARY OUTCOMES:
DLT | About 2 years
  Dose limiting toxicity
MTD | About 2 years
  Maximum tolerated dose

SECONDARY OUTCOMES:
Assessment of the safety after FLT3-targeted chimeric antigen receptor T cells infusion (Safety) | About 2 years
  Number of participants with treatment-related adverse events as assessed by CTCAE v5.0.
Assessment of pharmacokinetic (about Cmax) | About 28 days
  Assessment of the highest concentration (Cmax) of FLT3-targeted chimeric antigen receptor T cells amplified in peripheral blood after administration.
Assessment of pharmacokinetic (about Tmax) | About 28 days
  Assessment of the time to reach the highest concentration (Tmax) of FLT3-targeted chimeric antigen receptor T cells amplified in peripheral blood after administration.
Assessment of pharmacokinetic (about AUC0-28d) | About 28 days
  Assessment of the area under the curve AUC0-28d after administration.
Assessment of pharmacokinetic (about AUC0-90d) | About 90 days
  Assessment of the area under the curve AUC0-90d after administration. Assessment of the area under the curve AUC0-90d after administration. Assessment of the area under the curve AUC0-90d after administration.
PD endpoints | About 2 years
  The proportion and absolute value of FLT3-positive cells in peripheral blood at each time point; concentration levels of CAR-T-related serum cytokines such as CRP and IL-6.
To Evaluate Anti-tumour Activity (overall response rate) | About 3 months
  Rate of participants who with lymphoma aquire complete response (CR) or partial response (PR) or those who with leukemia CR or CR with incomplete hematologic recovery (CRi).
To Evaluate Anti-tumour Activity (Overall Survival) | About 2 years
  Defined as the time from start of FLT3 CAR-T cell therapy to death (due to any cause)
To Evaluate Anti-tumour Activity (duration of response) | About 2 years
  Defined as the time from the first tumor assessment of CR or PR , CR or CRi to the first assessment of disease recurrence or progression or death (due to any cause).
To Evaluate Anti-tumour Activity (Progression Free Survival) | About 2 years
  Defined as the time from the start of FLT3 CAR-T cell therapy to the first disease progression or recurrence or death from any cause.
Immunogenicity endpoints | About 2 years
  Positive rate of human anti-CAR antibody at each time point.

CONTACTS AND LOCATIONS:
Overall Officials: Heng Mei, MD, Principal Investigator — Union Hospital, Tongji Medical College, Huazhong University of Science and Technology
Locations (1):
- Union Hospital, affiliated with TongJi Medical College, HuaZhong University of Science and Technology, Wuhan, Hubei, China